CLINICAL TRIAL: NCT00877825
Title: The Influence of Soy Isoflavnoids on the Hypocholesterolemic Effects of Soy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REB235U
Record Dates: First submitted 2009-04-03; First posted 2009-04-08 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Hyperlipidemia; Cardiovascular Diseases
Keywords: Diet Therapy
MeSH Terms: conditions — Hyperlipidemias; Cardiovascular Diseases

INTERVENTIONS:
Procedure: dairy food control diet and high- and low- isoflavone soyfood diets

SUMMARY:
Isoflavonoids, through their estrogen-like activity, are in part responsible for the cholesterol lowering properties of soy foods. If this is found to be so, then it would be advantageous not only to promote soy consumption, but also to identify and use soy cultivars with high isoflavonoid content in production of soy food products. These foods may have a use in the reduction of serum cholesterol and if they effectively increase the phytoestrogen activity of soy, may have a role in the prevention of other hormone dependent diseases (e.g. osteoporosis, certain cancers) in the same way as natural estrogens.

ELIGIBILITY:
Inclusion Criteria:

* men and post-menopausal women
* LDL-C > 4.1mmol/L at recruitment
* living within a 40 km radius of St. Michael's Hospital

Exclusion Criteria:

* lipid lowering medications
* clinical or biochemical evidence of diabetes, renal or hepatic disease
* body mass index (BMI) >38 kg/m2
* antibiotic use within the last three months
* hormone replacement therapy
* smoking or significant alcohol use (>1 drink/d)
* triglyceride level > 4.0mmol/L

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Study Completion 2000-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David JA Jenkins, MD, PhD, DSc, Principal Investigator — University of Toronto and St. Michael's Hospital

REFERENCES:
- [Derived] Wong JM, Kendall CW, Marchie A, Liu Z, Vidgen E, Holmes C, Jackson CJ, Josse RG, Pencharz PB, Rao AV, Vuksan V, Singer W, Jenkins DJ. Equol status and blood lipid profile in hyperlipidemia after consumption of diets containing soy foods. Am J Clin Nutr. 2012 Mar;95(3):564-71. doi: 10.3945/ajcn.111.017418. Epub 2012 Feb 1. PMID 22301925